CLINICAL TRIAL: NCT01557062
Title: Passive Body Heating Improves The Sleep Pattern In Women Patients Fibromyalgia
Brief Title: Passive Body Heating, Sleep and Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Marco Tulio de Mello, Ph.D, Federal University of São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fibromyalgia_0866/06
Record Dates: First submitted 2012-03-09; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Hydrotherapy; Sleep; Pain; Body Temperature
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Polysomnography (Other)
  Interventions: Other: Polysomnography
- Temperature measure (Other)
  Interventions: Other: Teperature measure
- Fibromyalgia Impact questionary (Other)
  Interventions: Other: Fibromyalgia Impact questionary

INTERVENTIONS:
Other: Polysomnography — The Embla® S7000 was used to record full-night at the Sleep Institute (São Paulo, Brazil). The sensors were attached to the patient in a non-invasive manner using tape or rubber bands. The physiological variables were monitored simultaneously and continuously: 4 channels of EEG, 2 of EOG, 4 of EMG and 1 channel of ECG. Airflow detection was made through 2 channels using a pair of thermal sensors and nasal pressure. Respiratory effort of the chest and abdomen, were measured by respiratory inductance plethysmography. Oxygen saturation, were measured with a pulse oximeter. Sleep stages were visually scored in all the PSG according to standardized criteria for the investigation of sleep macrostructure.
  Arms: Polysomnography
Other: Teperature measure — Core body temperature was assessed using a thermistor pill (sensor), which is an electronic device 2.23 cm in length and 1.06 cm in diameter that records body temperature and transmits it to a receptor located at the patient's waist called the Core Body Temperature Monitoring System (CorTempTM), that is powered by a silver oxide battery. The components of the sensor are encapsulated in epoxy resin and coated with silicone (HQ Inc., Florida, USA). To ensure that the sensor would be in the intestines and not the stomach, the pill was ingested at least 2 hours (h) before beginning temperature recording. The CBT was recorded every 30 minutes (min) between 10:00pm and 7:00am. The time of pill elimination is variable between individuals and may be as long as 48h.
  Arms: Temperature measure
Other: Fibromyalgia Impact questionary — The FIQ is an instrument used to assess the quality of life specifically for patients with FM. This questionnaire consists of 19 questions related to functional capacity, employment status, general well being, psychological disorders and physical symptoms. The higher the score is, the greater is the impact of FM in the individual's quality of life. This questionnaire was validated for Brazilian's population in 2006.
  Arms: Fibromyalgia Impact questionary

SUMMARY:
Objectives: To assess the effect of passive body heating on the sleep pattern of patients with fibromyalgia.

Methods: Six menopausal women diagnosed with fibromyalgia according to criteria determined by the American College of Rheumatology were included. All women underwent passive immersion in a warm bath at 36±1 °C, for 15 sessions of 30 minutes each over 3 weeks. Their sleep pattern was assessed by polysomnography at the following conditions: pre-intervention (baseline), on the first day of intervention (acute), on the last day of intervention (chronic) and 3 weeks after the end of interventions (follow-up). Core body temperature was evaluated by a thermistor pill at the above-mentioned conditions. The impact on fibromyalgia was assessed through of a specific questionnaire called fibromyalgia impact questionnaire.

DETAILED DESCRIPTION:
Patients were attended at the Psychobiology and Exercise Studies Centre 5 times a week for 3 weeks between 6:00pm and 8:00pm for passive body-heating interventions for 30 min each session. The patients were accompanied by a researcher to a therapeutic water bath (Barritz Hydrotherapy Appliance, Germany) and were comfortably positioned in a supine position with their necks supported by an inflatable floating pillow to keep the body relaxed and safe during the intervention. The room temperature at the laboratory was maintained at 23±1 ºC, and the water temperature was 36±1ºC.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnostic
* Women
* Post menopausal
* Sedentary

Exclusion Criteria:

* Other diagnosis of chronic illnesses

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Sleep Pattern | 7 weeks. Was measured the sleep parameters from: Baseline to acute's time point (at the first day of intervention); Acute to chronic's time point (after 15 sections); Chronic's to follow-up time point (at 15 days after end point of interventions).
  Polysomnographies's register

SECONDARY OUTCOMES:
Impact of Fibromyalgia Disease | 7 weeks- The measurements occurred at the following time points: baseline, chronic and follow-up.
  Fibromyalgia Impact Questionnaire (FIQ)
Changes in Core Body Temperature (CBT) | 7 weeks. Was measured the CBT from: Baseline to acute's time point (at the first day of intervention); Acute to chronic's time point (after 15 sections); Chronic's to follow-up time point (at 15 days after end point of interventions).
  was monitored continuously throughout the nights at baseline and on days of the experimental protocols by a thermistor pill with a CorTemp HT150002 and core temperature sensor coupled with a data recorder.

CONTACTS AND LOCATIONS:
Overall Officials: Marco T De Mello, Ph.D, Principal Investigator — Federal University of São Paulo; Adressa Silva, MD, Study Chair — Federal University of São Paulo; Sandra S Queiroz, Study Chair — Federal University of São Paulo; Mônica L Andersen, Ph.D, Study Chair — Federal University of São Paulo; Marcos Mônico-Neto, Study Chair — Federal University of São Paulo; Raquel MS Campos, MD, Study Chair — Federal University of São Paulo; Suely Roizenblatt, Ph.D, Study Chair — Federal University of São Paulo; Sergio Tufik, Ph.D, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Vitorino DF, Carvalho LB, Prado GF. Hydrotherapy and conventional physiotherapy improve total sleep time and quality of life of fibromyalgia patients: randomized clinical trial. Sleep Med. 2006 Apr;7(3):293-6. doi: 10.1016/j.sleep.2005.09.002. Epub 2006 Mar 24. PMID 16564209
- [Background] Langhorst J, Musial F, Klose P, Hauser W. Efficacy of hydrotherapy in fibromyalgia syndrome--a meta-analysis of randomized controlled clinical trials. Rheumatology (Oxford). 2009 Sep;48(9):1155-9. doi: 10.1093/rheumatology/kep182. Epub 2009 Jul 16. PMID 19608724
- [Background] Evcik D, Kizilay B, Gokcen E. The effects of balneotherapy on fibromyalgia patients. Rheumatol Int. 2002 Jun;22(2):56-9. doi: 10.1007/s00296-002-0189-8. Epub 2002 Mar 29. PMID 12070676
- [Background] Bunnell DE, Agnew JA, Horvath SM, Jopson L, Wills M. Passive body heating and sleep: influence of proximity to sleep. Sleep. 1988 Apr;11(2):210-9. doi: 10.1093/sleep/11.2.210. PMID 3381061
- [Background] Jordan J, Montgomery I, Trinder J. The effect of afternoon body heating on body temperature and slow wave sleep. Psychophysiology. 1990 Sep;27(5):560-6. doi: 10.1111/j.1469-8986.1990.tb01976.x. PMID 2274619